CLINICAL TRIAL: NCT05389046
Title: Study on the Optimal Diagnosis and Treatment Strategy of Major Depressive Disorder Based on Anhedonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Si Tianmei, Professor, Peking University Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1-4111
Record Dates: First submitted 2022-05-15; First posted 2022-05-24 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Outpatients / Inpatients With Depression
Keywords: major depressive disorder; anhedonia; inflammatory immune; reward system; optimal treatment; neurotransmitter
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Escitalopram (Experimental): Escitalopram monotherapy (10-20 mg/day）
  Interventions: Drug: Escitalopram
- Escitalopram + omega-3 PUFAs (Experimental): Escitalopram (10-20 mg/day）combined with omega-3 PUFAs （EPA 900mg，DHA 300 mg）
  Interventions: Drug: Escitalopram+omega-3 PUFAs
- Escitalopram + Aripiprazole (Experimental): Escitalopram (10-20 mg/day）combined with Aripiprazole （2.5-10 mg/day)
  Interventions: Drug: Escitalopram+Aripiprazole
- Escitalopram + omega-3 PUFAs + Aripiprazole (Experimental): Escitalopram (10-20 mg/day）combined with omega-3 PUFAs （EPA 900mg，DHA 300 mg）and Aripiprazole （2.5-10 mg/day)
  Interventions: Drug: Escitalopram+Aripiprazole+omega-3 PUFAs

INTERVENTIONS:
Drug: Escitalopram — Escitalopram
  Arms: Escitalopram
Drug: Escitalopram+Aripiprazole — Escitalopram+Aripiprazole
  Arms: Escitalopram + Aripiprazole
Drug: Escitalopram+omega-3 PUFAs — Escitalopram+omega-3 PUFAs
  Arms: Escitalopram + omega-3 PUFAs
Drug: Escitalopram+Aripiprazole+omega-3 PUFAs — Escitalopram+Aripiprazole+omega-3 PUFAs
  Arms: Escitalopram + omega-3 PUFAs + Aripiprazole

SUMMARY:
This study is a multicenter clinical research and focuses on the exploring of optimal diagnosis and treatment strategies of MDD based on anhedonia.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a heterogeneious psychiatric disorder with complex etiology and pathogenesis. The lack of objective criteria for diagnosis and the use of trial-and-error treatment strategy are the current challenge. Anhedonia is the core symptom of MDD and the aberrant reward system and abnormal inflammatory immune may be the pathological mechanisms. Previous evidence suggests anhedonia cannot be improved quickly and efficiently by taking the first-line antidepressants. This study focuses on exploring the optimal diagnosis and treatment strategy for MDD patients with anhedonia. Based on the hypothesis of inflammatory-immune system，neurotransmitter abnormalities and aberrant reward system, this study aims to evaluate the efficacy and safety of the combinations of escitalopram and aripiprazole and/or omega-3 polyunsaturated fatty acids for MDD patients with anhedonia with a factorial design. Moreover, the multidimensional data including the clinicopathological features, neuroimaging data (MRI) and inflammatory cytokines will be used to establish the model of diagnosis and treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Major depressive disorder according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5);
2. Age: 18-55 (including 18 and 55)
3. HAMD-17≥18
4. DARS ≤ 28
5. Do not receive repetitive Transcranial Magnetic Stimulation (rTMS) or modified electroconvulsive therapy (MECT) treatment in past six months.
6. Sign the informed consent form voluntarily and agree to participate in all visits, examinations and treatment as required by the trial protocol.

Exclusion Criteria:

1. Patients who are diagnosed with major somatic diseases;
2. Patients who meet DSM-5 diagnostic criteria for other mental disorders: Personality disorder, mental retardation; drug and/or alcohol dependence;
3. Patients with severe suicidal tendencies or suicidal behavior;
4. Pregnant or lactating women;
5. Patients with MRI contraindications;
6. Patients who are regarded as unsuitable by investigators for this clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
17-item Hamilton depression rating scale (HAMD-17) value | Day 0 to Day 56
  The value of 17-item Hamilton depression rating scale (HAMD-17) total score treatment compared to that at the baseline. The maximum score of HAMD-17 is 51 and the minimum is 0. Higher scores mean a worse outcome.
Anhedonia level-Dimensional Anhedonia Rating Scale (DARS) | Day 0 to Day 56
  The outcome is measured by Dimensional Anhedonia Rating Scale (DARS) total score. The maximum score of DARS total score is 68 and the minimum is 0. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Anxiety symptoms | Day 0 to Day 14, Day 0 to Day 28, Day 0 to Day 56
  The outcome is measured by Hamilton anxiety rating scale (HAMA) total score change. The change value of HAMA total scores at each timepoints compared to the baseline. The maximum score of HAMA is 56 and the minimum is 0. Higher scores mean a worse outcome.

OTHER OUTCOMES:
cognition outcome | Day 0 to Day 56
  The outcome is measured by cognition task.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Xicheng District Pingan Hosptial, Beijing, Beijing Municipality
  - Beijing Huilongguan Hospital, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No